CLINICAL TRIAL: NCT02431273
Title: Open-Label Safety and Pharmacokinetic Study of Single (TDF), Dual (TDF-FTC), and Triple ARV IVR (TDF-FTC-MVC) in Healthy Women
Brief Title: Safety and Pharmacokinetic Study of HIV Prophylaxis Using Antiretroviral Intravaginal Rings in Healthy Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Auritec Pharmaceuticals (Industry)
Collaborators: The University of Texas Medical Branch, Galveston (Other); Oak Crest Institute of Science (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ARV-IVR 01; 2R44HD075636-02 (NIH)
Record Dates: First submitted 2014-08-04; First posted 2015-05-01 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Human Immunodeficiency Virus (HIV) Prophylaxis
Keywords: TDF; FTC; MVC; TDF-FTC; TDF-FTC-MVC; IVR; ARV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TDF (Single IVR) (Experimental): All subjects will be asked to wear "Single" (TDF) IVRs for 7 days.
  Interventions: Drug: TDF IVR
- TDF-FTC (Dual IVR) (Experimental): If the TDF IVR is determined as safe, study participants will be asked to replace it with "Dual" (TDF-FTC) IVRs for 7 days. There will be follow-up visit between removal of a single IVR and replacing it with a dual IVR.
  Interventions: Drug: TDF-FTC IVR
- TDF-FTC-MVC (Triple IVR) (Experimental): If the TDF-FTC IVR is determined as safe, study participants will be asked to replace them with "Triple" (TDF-FTC-MVC) IVRs for 7 days. There will be follow-up visit between removal of a dual IVR and replacing it with a triple IVR.
  Interventions: Drug: TDF-FTC-MVC IVR

INTERVENTIONS:
Drug: TDF IVR
  Other Names: Single IVR
  Arms: TDF (Single IVR)
Drug: TDF-FTC IVR
  Other Names: Dual IVR
  Arms: TDF-FTC (Dual IVR)
Drug: TDF-FTC-MVC IVR
  Other Names: Triple IVR
  Arms: TDF-FTC-MVC (Triple IVR)

SUMMARY:
This study will evaluate the hypothesis that intravaginal rings (IVRs) can safely and in a sustained fashion, deliver the antiretroviral (ARV) drugs - tenofovir disoproxil fumarate (TDF), emtricitabine (FTC), and maraviroc (MVC), in healthy women when used in the following drug combinations: 1) TDF ("Single" IVR); 2) TDF-FTC ("Dual" IVR) and; 3) TDF-FTC-MVC ("Triple" IVR).

TDF = tenofovir disoproxil fumarate; FTC = emtrcitabine; MVC = maraviroc

DETAILED DESCRIPTION:
The broad long term goal of this project is to empower women to protect themselves from HIV through woman-controlled sustained local delivery of ARTs via intravaginal rings. The short-term general investigational plan is to evaluate IVRs releasing TDF, TDF-FTC and TDF-FTC-MVC in healthy women for up to 7 days in an open-label study to determine safety and drug concentrations in plasma and cervicovaginal lavage and secretions. Additional exploratory studies will be considered and planned based in part on the results obtained in this study. The long-term investigational plan is to evaluate the safety and efficacy of sustained release TDF, TDF-FTC and TDF-FTC-MVC for their ability to decrease HIV transmission to vulnerable women.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Healthy female 18-45 years of age
* HIV negative per subject report and results of screening examination
* Negative for sexually transmitted diseases in the past 3 months and at screening exam
* No history of genital herpes simplex I or II per subject report
* Currently using contraception with plans to continue throughout the study duration or having sex with females only
* Pre-menopausal with a regular menstrual cycle with at least 21 days between menses and no history of intermenstrual bleeding or with suppressed menstrual cycle by hormonal contraception such as Depo-Provera or continuous oral contraceptive agents
* Subjects must agree to abstain from vaginal, anal, and oral sex throughout the first week of each dosing period and then use condoms for vaginal/rectal intercourse until after the final visit for use of each IVR
* Subjects must agree to not douche or use any vaginal product other than the Single, Dual and Triple ARV IVRs, including lubricants, feminine hygiene products, and vaginal drying agents throughout the dosing period and until after the final visit
* Subjects must agree to blood draws and vaginal exams throughout the course of the study

Exclusion Criteria:

* HIV positive by subject report or results of screening examination
* Positive history for autoimmune disease
* Abnormal genital exam defined as grade 1 or higher adverse event by DAIDS genital AE grading table
* Abnormal ALT or AST or Hepatitis B infection
* Active vaginal infection as determined by site IoR
* Abnormal renal function (defined as a creatinine clearance of <50mL/min/1.73 m2)
* Pregnant or less than 6 months post-partum or current lactation
* Current use of an IVR (i.e., Nuvaring, Estring, Femring)
* History of TDF, FTC, and MVC use and/or adverse reaction to any of these drugs
* History of adverse reaction to silicone
* History of toxic shock syndrome
* Currently receiving chemotherapy or immunosuppressive agents
* Use of investigative drugs within 30 days or 5 half-lives
* Currently using or suspected to be using non-therapeutic injection drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Vincent, MD, Principal Investigator — University of Texas Medical Branch (UTMB)
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Vincent KL, Moss JA, Marzinke MA, Hendrix CW, Anton PA, Pyles RB, Guthrie KM, Dawson L, Olive TJ, Butkyavichene I, Churchman SA, Cortez JM Jr, Fanter R, Gunawardana M, Miller CS, Yang F, Rosen RK, Vargas SE, Baum MM. Safety and pharmacokinetics of single, dual, and triple antiretroviral drug formulations delivered by pod-intravaginal rings designed for HIV-1 prevention: A Phase I trial. PLoS Med. 2018 Sep 28;15(9):e1002655. doi: 10.1371/journal.pmed.1002655. eCollection 2018 Sep. PMID 30265679
- [Derived] Moss JA, Butkyavichene I, Churchman SA, Gunawardana M, Fanter R, Miller CS, Yang F, Easley JT, Marzinke MA, Hendrix CW, Smith TJ, Baum MM. Combination Pod-Intravaginal Ring Delivers Antiretroviral Agents for HIV Prophylaxis: Pharmacokinetic Evaluation in an Ovine Model. Antimicrob Agents Chemother. 2016 May 23;60(6):3759-66. doi: 10.1128/AAC.00391-16. Print 2016 Jun. PMID 27067321

RESULTS

PARTICIPANT FLOW:
Groups:
- TDF (Single IVR), TDF-FTC (Dual IVR), TDF-FTC-MVC (Triple IVR): All subjects will be asked to wear TDF (Single) IVRs for 7 days.
  If the TDF IVR is determined as safe, study participants will be asked to replace it with "Dual" (TDF-FTC) IVRs for 7 days.
  If the TDF-FTC IVR is determined as safe, study participants will be asked to replace them with "Triple" (TDF-FTC-MVC) IVRs for 7 days.
Period: TDF (Single IVR)
Arm/Group | TDF (Single IVR), TDF-FTC (Dual IVR), TDF-FTC-MVC (Triple IVR)
Started | 6
Completed (All 6 participants that completed Period 1 (TDF IVR) screened for Period 2 (TDF-FTC IVR)) | 6
Not Completed | 0
Period: TDF-FTC (Dual IVR)
Arm/Group | TDF (Single IVR), TDF-FTC (Dual IVR), TDF-FTC-MVC (Triple IVR)
Started | 6
Completed (2 of 6 participants that completed Period 2 (TDF-FTC IVR) screened for Period 3 (TDF-FTC-MVC IVR)) | 6
Not Completed | 0
Period: TDF-FTC-MVC (Triple IVR)
Arm/Group | TDF (Single IVR), TDF-FTC (Dual IVR), TDF-FTC-MVC (Triple IVR)
Started | 6
Completed (2 participants that completed Periods 1 and 2, along with 4 new subjects participated in Period 3) | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 6 subjects were screened, entered, and completed Period 1: TDF-IVR (Single IVR).
  The 6 subjects then completed Period 2: TDF-FTC (Dual IVR). 4 of the 6 subjects dropped out afterward.
  2 of the 6 original subjects, plus 4 new subjects entered Period 3: TDF-FTC-MVC (Triple IVR).
  Here, baseline data of all subjects are presented.
Groups:
- All Study Participants: All subjects will be asked to wear "Single" (TDF) IVRs for 7 days.
  If the TDF IVR is determined as safe, study participants will be asked to replace it with "Dual" (TDF-FTC) IVRs for 7 days. There will be follow-up visit between removal of a single IVR and replacing it with a dual IVR.
  If the TDF-FTC IVR is determined as safe, study participants will be asked to replace them with "Triple" (TDF-FTC-MVC) IVRs for 7 days. There will be follow-up visit between removal of a dual IVR and replacing it with a triple IVR.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] — Population: 6 subjects were screened, entered, and completed Period 1: TDF-IVR (Single IVR) and Period 2: TDF-FTC (Dual IVR).
  2 of the 6 original subjects, plus 4 new subjects entered Period 3: TDF-FTC-MVC (Triple IVR). Total of 6 subjects were analyzed for each Period.
  years
    Period 1 and Period 2: number analyzed (Participants) | 6
    Period 1 and Period 2 | 26 [24 to 35]
    Period 3: number analyzed (Participants) | 6
    Period 3 | 24.5 [21 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Specific Graded Adverse Events in Single, Dual, and Triple Antiretroviral (ARV) Intravaginal Rings (IVRs)
Description: Number of Adverse Events (AEs) was recorded. Safety parameters were monitored for each IVR combination and the grading scale for each parameter followed the Female Genital Grading Table for Use in Microbicide Studies. AEs not included in that table were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 (Grade 1 = mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Potentially Life-Threatening).
Time Frame: Days 0-21 following insertion of each IVR.
Measure: Number; unit: participants
Groups:
- Period 1: TDF (Single IVR): All subjects will be asked to wear "Single" (TDF) IVRs for 7 days.
  TDF IVR
- Period 2: TDF-FTC (Dual IVR): If the TDF IVR is determined as safe, study participants will be asked to replace it with "Dual" (TDF-FTC) IVRs for 7 days. There will be follow-up visit between removal of a single IVR and replacing it with a dual IVR.
  TDF-FTC IVR
- Period 3: TDF-FTC-MVC (Triple IVR): If the TDF-FTC IVR is determined as safe, study participants will be asked to replace them with "Triple" (TDF-FTC-MVC) IVRs for 7 days. There will be follow-up visit between removal of a dual IVR and replacing it with a triple IVR.
  TDF-FTC-MVC IVR
Arm/Group | Period 1: TDF (Single IVR) | Period 2: TDF-FTC (Dual IVR) | Period 3: TDF-FTC-MVC (Triple IVR)
Number analyzed (Participants) | 6 | 6 | 6
participants
  Pelvic Pain: Grade 1 | 4 | 1 | 4
  Pelvic Pain: Grade 2 | 1 | 1 | 0
  Vaginal Discharge: Grade 1 | 3 | 3 | 1
  Metrorrhagia: Grade 1 | 1 | 0 | 2
  Vulvovaginal Itching: Grade 1 | 3 | 0 | 1
  Cervicovaginal Erythema: Grade 1 | 3 | 1 | 0
  Diarrhea: Grade 1 | 1 | 0 | 0
  Malaise: Grade 1 | 1 | 0 | 0
  Odor: Grade 1 | 0 | 0 | 1
  Nausea: Grade 1 | 0 | 0 | 1
  Candida (monilial vulvovaginitis): Grade 2 | 0 | 0 | 1

2. Primary Outcome: Pharmacokinetics of the Single, Dual and Triple ARV IVRs: Cervicovaginal Fluid (CVF)
Description: Drug concentrations [tenofovir (TFV), tenofovir disoproxil fumarate (TDF), emtricitabine (FTC) and maraviroc (MVC)] in cervicovaginal fluids (CVF) for each IVR combination.
Time Frame: Time points at which outcome measure was assessed are Days 2 (after IVR insertion) and 7 (day of IVR removal).
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | Period 1: TDF (Single IVR) | Period 2: TDF-FTC (Dual IVR) | Period 3: TDF-FTC-MVC (Triple IVR)
Number analyzed (Participants) | 6 | 6 | 6
ng/mg
  tenofovir disoproxil fumarate | 58.1 [43.9 to 97.4] | 43.1 [31.0 to 65.0] | 96.9 [14.5 to 137.1]
  tenofovir | 13.9 [6.2 to 19.3] | 15.9 [7.1 to 20.0] | 28.0 [24.3 to 31.9]
  Total tenofovir | 36.2 [31.3 to 60.6] | 34.4 [26.9 to 48.7] | 70.0 [59.2 to 80.6]
  emtricitabine | NA [NA to NA] — The IVR did not contain emtricitabine | 896 [367.0 to 1349.0] | 838.5 [641.8 to 1171.2]
  maraviroc | NA [NA to NA] — The IVR did not contain maraviroc | NA [NA to NA] — The IVR did not contain maraviroc | 429.8 [253.2 to 626.2]

3. Primary Outcome: Pharmacokinetics of the Single, Dual and Triple ARV IVRs: Cervicovaginal Lavage (CVL)
Description: Drug concentrations [tenofovir disoproxil fumarate (TDF), emtricitabine (FTC) and maraviroc (MVC)] in cervicovaginal lavage (CVL) were evaluated for each IVR combination.
Time Frame: Time points at which outcome measure was assessed are Days 2 (after IVR insertion) and 7 (day of IVR removal).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Period 1: TDF (Single IVR) | Period 2: TDF-FTC (Dual IVR) | Period 3: TDF-FTC-MVC (Triple IVR)
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  tenofovir disoproxil fumarate | 1,930 [1,040 to 2,290] | 1,720 [1,028 to 3,429] | 3,630 [2,310 to 15,700]
  tenofovir | 611 [242 to 2,440] | 927 [315 to 1,253] | 2,670 [1,668 to 4,175]

4. Primary Outcome: Pharmacokinetics of the Single, Dual and Triple ARV IVRs: Vaginal Tissue
Description: Drug concentrations [tenofovir disoproxil fumarate (TDF), tenofovir (TFV), tenofovir diphosphate (TFV-DP), emtricitabine (FTC) and maraviroc (MVC)] in vaginal tissue (VT) were evaluated for each IVR combination.
Time Frame: Time points at which outcome measure was assessed are Days 2 (after IVR insertion) and 7 (day of IVR removal).
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | Period 1: TDF (Single IVR) | Period 2: TDF-FTC (Dual IVR) | Period 3: TDF-FTC-MVC (Triple IVR)
Number analyzed (Participants) | 6 | 6 | 6
ng/mg
  tenofovir | 8.4 [4.7 to 11.2] | 5.1 [0.8 to 10.1] | 5.1 [3.3 to 9.7]
  tenofovir diphosphate | 303 [277 to 938] | 289 [110 to 603] | 301.9 [177.1 to 823.8]
  emtricitabine | NA [NA to NA] — The IVR did not contain emtricitabine | 23,950 [11,373 to 56,400] | 104 [63.7 to 301.7]
  maraviroc | NA [NA to NA] — The IVR did not contain maraviroc | NA [NA to NA] — The IVR did not contain maraviroc | 141.8 [82.5 to 212]

5. Primary Outcome: Pharmacokinetics of the Single, Dual and Triple ARV IVRs: Plasma
Description: Drug concentrations [tenofovir disoproxil fumarate (TDF), emtricitabine (FTC) and maraviroc (MVC)] in plasma were evaluated for each IVR combination.
Time Frame: Time points at which outcome measure was assessed are Days 2 (after IVR insertion) and 7 (day of IVR removal).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Period 1: TDF (Single IVR) | Period 2: TDF-FTC (Dual IVR) | Period 3: TDF-FTC-MVC (Triple IVR)
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  tenofovir: Plasma | NA [NA to NA] — Data is below the lower limit of quantification | NA [NA to NA] — Data is below the lower limit of quantification | NA [NA to NA] — Data is below the lower limit of quantification
  emtricitabine: Plasma | NA [NA to NA] — The IVR did not contain emtricitabine | 0.95 [0.91 to 1.14] | 1.02 [0.56 to 1.22]
  maraviroc: Plasma | NA [NA to NA] — The IVR did not contain maraviroc | NA [NA to NA] — The IVR did not contain maraviroc | 0.08 [0.05 to 0.14]

6. Primary Outcome: Pharmacokinetics of the Single, Dual and Triple ARV IVRs: Terminal Half-life
Description: Drug concentrations [tenofovir disoproxil fumarate (TDF), emtricitabine (FTC) and maraviroc (MVC)] in terminal half-life were evaluated for each IVR combination.
Time Frame: Time points at which outcome measure was assessed are Day 7 (day of IVR removal) and daily up to 14 days.
Measure: Median (Inter-Quartile Range); unit: Hour
Arm/Group | Period 1: TDF (Single IVR) | Period 2: TDF-FTC (Dual IVR) | Period 3: TDF-FTC-MVC (Triple IVR)
Number analyzed (Participants) | 6 | 6 | 6
Hour
  tenofovir disoproxil fumarate: Terminal Half-life | 11.8 [10.6 to 14.4] | 14.2 [11.7 to 15.4] | 18.3 [11.8 to 24.2]
  tenofovir: Terminal Half-life | 39.5 [30.0 to 58.1] | 31.4 [25.9 to 36.2] | 24.8 [24.4 to 31.9]
  emtricitabine: Terminal Half-life | NA [NA to NA] — The IVR did not contain emtricitabine | 19.1 [13.5 to 20.1] | 17.0 [15.5 to 17.8]
  maraviroc: Terminal Half-life | NA [NA to NA] — The IVR did not contain maraviroc | NA [NA to NA] — The IVR did not contain maraviroc | 16.0 [15.8 to 18.3]

7. Secondary Outcome: Acceptability of the IVRs
Description: Acceptability of the IVRs was assessed through reported willingness to use the IVR for 28 days in a real-world setting on a likert scale, 1 being "not at all confident" to 5 being "completely confident" for Periods 1 and 2.
Time Frame: Days 0-21 following insertion of each IVR.
Population: Data was not collected for the third study period.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Period 1: TDF (Single IVR) | Period 2: TDF-FTC (Dual IVR) | Period 3: TDF-FTC-MVC (Triple IVR)
Number analyzed (Participants) | 6 | 6 | 0
units on a scale | 3.5 [1 to 5] | 4 [1 to 5] |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected Days 0-21 following insertion of each IVR. Safety measures include: daily participant reports, colposcopy examinations, vaginal microbiome evaluations, or histology from vaginal biopsy.
Groups:
- TDF (Single IVR): All subjects will be asked to wear "Single" (TDF) IVRs for 7 days.
  TDF IVR
- TDF-FTC (Dual IVR): If the TDF IVR is determined as safe, study participants will be asked to replace it with "Dual" (TDF-FTC) IVRs for 7 days. There will be follow-up visit between removal of a single IVR and replacing it with a dual IVR.
  TDF-FTC IVR
- TDF-FTC-MVC (Triple IVR): If the TDF-FTC IVR is determined as safe, study participants will be asked to replace them with "Triple" (TDF-FTC-MVC) IVRs for 7 days. There will be follow-up visit between removal of a dual IVR and replacing it with a triple IVR.
  TDF-FTC-MVC IVR
Arm/Group | TDF (Single IVR) | TDF-FTC (Dual IVR) | TDF-FTC-MVC (Triple IVR)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF (Single IVR) (N=6) | TDF-FTC (Dual IVR) (N=6) | TDF-FTC-MVC (Triple IVR) (N=6)
Pelvic Pain (Reproductive system and breast disorders) | 3 (5) | 2 (3) | 4 (5) — Relationship: Possibly Related
Vaginal Discharge (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 1 (1) — Relationship: Possibly Related
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) — Relationship: Possibly Related
Vulvovaginal Itching (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 1 (1) — Relationship: Possibly Related
Cervicovaginal Erythema (Reproductive system and breast disorders) | 3 (3) | 1 (3) | 0 (0) — Relationship: Possibly Related
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Relationship: Possibly Related
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) — Relationship: Not Related
Odor (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Relationship: Possibly Related
Nausea (General disorders) | 0 (0) | 0 (0) | 1 (1) — Relationship: Possibly Related
Candida (monilial vulvovaginitis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Relationship: Possibly Related

LIMITATIONS AND CAVEATS:
The study's main limitations include the small sample size, short duration (7 days), and the lack of FTC triphosphate measurements in vaginal tissue biopsies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No